CLINICAL TRIAL: NCT00319579
Title: The Long Term Medical and Psychological Implications of Becoming a Living Kidney Donor: A Prospective Pilot Study
Brief Title: Pilot Prospective Study: Long-term Health of Living Kidney Donors
Status: Completed | Type: Observational
Sponsor: Amit Garg (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Amit Garg, MD, MA, FRCPC, FACP, PhD, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Other Study IDs: R-04-204; LKD Prospective Study
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Living Kidney Donors
Keywords: living kidney donors; prospective; medical; psychosocial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Living Kidney Donors with controls who have not donated a kidney and meet certain criteria at the time of the donor's donation (i.e. no hypertension, no kidney disease, etc.).

SUMMARY:
Kidney transplantation, a 'miracle' of modern medicine, is the preferred treatment option for End Stage Renal Disease compared to dialysis, patients who receive kidneys have a 70% reduction in risk of death, a dramatically improved quality of life and cost the health care system considerably less. As a result there are over 3000 Canadians, and 57,000 Americans on the waiting list for a kidney. To meet the shortage in cadaveric kidneys, rates of living kidney donation have nearly doubled over the last 10 years, and will continue to rise with growing demand.

Yet despite its advantages for the recipient, living kidney donation remains a complex ethical, moral and medical issue. The premise for accepting living donors is that the "minimal" risk of short and long-term medical harm realized by the donor is outweighed by the definite advantages to the recipient and potential psychosocial benefits of the altruistic gift to the donor. The only benefit for the living donor is psychological - donors experience increased self-esteem, feelings of well-being and improved health related quality of life with their altruistic act of assuming medical risk to help another. The short-term consequences of living donation are well established. On the other hand the long-term implications of living kidney donation are far less certain. This study will look at the long term implications of living kidney donation.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years old
2. A predicted Cockcroft-Gault creatinine clearance > 80 mL/min
3. Average sBP < 140 and dBP < 90 based on 3 readings
4. A spot urine protein to creatinine ratio < 15 mg/mmol

Exclusion Criteria:

1. A medical condition (such as cardiovascular disease, pulmonary disease, active cancer) or psychological condition (such as major affective disorder, personality disorder, a history of chemical dependence) which the local transplant centre deems unfit for donation. Blood group and immunological incompatibility (such as positive cross-match, poor HLA matches) are not reasons for exclusion
2. Evidence of a financial incentive for donation
3. A contraindication to general anaesthesia or surgery
4. A past medical history of hypertension
5. Use of antihypertensive class medications for any reason.(ACE-Is, ARBs, diuretics, beta-blockers, calcium channel blockers)
6. A past history of permanent proteinuria
7. The eligible non-donor is planning to donate their kidney within the next year
8. Unable to give informed consent
9. Unwilling to participate in the follow-up assessments at one, two, three, four and five years, or unwilling or unable to conduct home blood pressure or laboratory measurements
10. The living donor or eligible non-donor is currently pregnant
11. Despite being planned the donor nephrectomy does not take place
12. Enrolled in another clinical study which interferes with the conduct or outcomes of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Living Kidney Donors
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Hypertension in living kidney donors | Annually for 5 years post donation

CONTACTS AND LOCATIONS:
Overall Officials: Amit X Garg, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (15):
- United States (5):
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Yale University and VAMC, West Haven, Connecticut
  - Wayne State University, Detroit, Michigan
  - Cleveland Clinic, Cleveland, Ohio
  - Hume-Lee Transplant Center Renal/Pancreas Transplant Program, Richmond, Virginia
- Australia (2):
  - MonashMedical Centre, Clayton, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Canada (8):
  - University of Alberta, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Dalhousie University, Halifax, Nova Scotia
  - St. Joseph Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Garcia-Ochoa C, Feldman LS, Nguan C, Monroy-Caudros M, Arnold JB, Barnieh L, Boudville N, Cuerden MS, Dipchand C, Gill JS, Karpinski M, Klarenbach S, Knoll G, Lok CE, Miller M, Prasad GVR, Sontrop JM, Storsley L, Garg AX. Impact of Perioperative Complications on Living Kidney Donor Health-Related Quality of Life and Mental Health: Results From a Prospective Cohort Study. Can J Kidney Health Dis. 2021 Aug 11;8:20543581211037429. doi: 10.1177/20543581211037429. eCollection 2021. PMID 34394947
- [Derived] Garcia-Ochoa C, Feldman LS, Nguan C, Monroy-Cuadros M, Arnold J, Boudville N, Cuerden M, Dipchand C, Eng M, Gill J, Gourlay W, Karpinski M, Klarenbach S, Knoll G, Lentine KL, Lok CE, Luke P, Prasad GVR, Sener A, Sontrop JM, Storsley L, Treleaven D, Garg AX; Donor Nephrectomy Outcomes Research (DONOR) Network. Perioperative Complications During Living Donor Nephrectomy: Results From a Multicenter Cohort Study. Can J Kidney Health Dis. 2019 Jul 18;6:2054358119857718. doi: 10.1177/2054358119857718. eCollection 2019. PMID 31367455